CLINICAL TRIAL: NCT05768750
Title: A Home-based Rehabilitation Program to Counter the Motor Impairments and Activity Limitations Experienced by People With Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay
Brief Title: A Home-based Rehabilitation in ARSACS
Acronym: PACE-ARSCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Cynthia Gagnon, Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-047
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Autosomal Recessive Spastic Ataxia of Charlevoix-Saguenay
Keywords: ARSACS
MeSH Terms: conditions — Spastic ataxia Charlevoix-Saguenay type | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will participate in 2 phases : control phase (12-week usual care) followed by an intervention phase (12-week home-based rehabilitation program).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control followed by intervention phase (Experimental): All participants will participate in 2 phases : control phase (12-week usual care) followed by an intervention phase (12-week home-based rehabilitation program).
  The rehabilitation program consists of three domains of exercises divided by levels of difficulty: sitting balance (16 levels), standing balance (21 levels) and sit-to-stand transfer (12 levels), including 67 exercises. Each individualized home-based rehabilitation program will include 3 to 6 exercises, for a total duration of 15 to 20 minutes.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — X

SUMMARY:
48 participants (24 women and 24 men) with autosomal recessive spastic ataxia of Charlevoix-Saguenay (ARSACS) will participate in 2 phases : control phase (12-week usual care) and intervention phase (12-week home-based rehabilitation program). The participants will be evaluated at baseline, week 12 (end of control phase) and week 24 (end of intervention phase) to quantify the effects of an individualized home-based rehabilitation program. Participants will also participate on a focus group at the end of the program to evaluate the acceptability of the program and the perceived changes.

DETAILED DESCRIPTION:
Co-creation phase:

Preceding the intervention, a co-creation phase involving healthcare professionals (3), patient-partners (2), and ARSACS researchers (3) will be conducted to develop the exercises for the rehabilitation program and the evaluation scale to determine the level of difficulty of each exercise assigned to participants.

Intervention phase:

Random sampling stratified by gender and level of indoor mobility (unassisted walking, assisted walking, wheelchair) from the Neuromuscular Clinic's registry of 48 participants (24 women and 24 men) will be conducted.

* Control phase: All participants will be asked to maintain their usual activities for 12 weeks.
* Intervention phase: All participants recruited to the project will complete the home-based rehabilitation program assigned to them for 12 weeks, unsupervised, 20 minutes 3 times a week. Follow-up calls by a physiotherapist will be conducted at weeks 2, 4, 6, 8, 10 and 12.

ELIGIBILITY:
Inclusion Criteria:

* ARSACS diagnosis must be confirmed by genetic analysis;
* Women and men, aged between 18 and 50 years old;
* Be able to perform the sit-to-stand transfer;
* Consent of the neurologist must be given to participate in this study;
* Must reside in the Saguenay-Lac-St-Jean region;
* Subjects must be able to give their consent freely and voluntarily.

Exclusion Criteria:

* Patients who already meet physical activity (PA) recommendations (150 min of moderate to high intensity PA/week) or already participate in a rehabilitation program are excluded;
* Remain in a care facility;
* Do not speak English or French;
* Have another diagnosis causing physical limitations;
* Are pregnant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in sitting balance | Baseline, week 12, week 24
  Measured with the Ottawa sitting scale, score range 0-40, a higher score indicates a better outcome
Change in balance | Baseline, week 12, week 24
  Measured with the Berg Balance Scale, score range 0-56, a higher score indicates better balance
Change in walking speed | Baseline, week 12, week 24
  Change in the walking speed, measured with the time to walk 10 meters at self-selected and maximum speed

SECONDARY OUTCOMES:
Change in the balance confidence | Baseline, week 12, week 24
  Measured with the modified Activities-specific Balance Confidence (ABC) Scale, score range 0-100, 0 indicates no confidence and 100 is full confidence
Change in the number of falls | Baseline, week 12, week 24
  Number of self-reported falls in the last month
Change in the lower limb coordination | Baseline, week 12, week 24
  Number of touched targets in a 30 second period with each foot, measured with the Lower Extremity MOtor COordination Test (LEMOCOT)
Change in the number of sit-to-stand performed in 30 seconds | Baseline, week 12, week 24
  Number of complete sit-to-stand performed in 30 seconds without the help of arms
Change in the time required to ascent 10 stairs | Baseline, week 12, week 24
  Time required to ascent 10 stairs, measured with the 10 Stairs Ascent
Change in the time required to descent 10 stairs | Baseline, week 12, week 24
  Time required to descent 10 stairs, measured with the 10 Stairs Descent
Change in the life space | Baseline, week 12, week 24
  Measured with the Life Space Assessment (LSA), score range 0-120, a higher score indicates higher level of mobility in the next five areas: outside the bedroom, outside the house, in the neighborhood, outside of the neighborhood but in town, and outside town during the past four weeks
Change in the upper limb coordination | Baseline, week 12, week 24
  Number of finger touched targets in a 20 second period of each side, measured with the Standardized Finger-Nose Test (SFNT)
Change in social participation | Baseline, week 12, week 24
  The performance in activities of daily living, measured with the Assessment of Life Habits (LIFE-H), score range 0-9
Change in the Scale for the assessement and rating of ataxia (SARA) | Baseline, week 12, week 24
  Measured with the Scale for the assessment and rating of ataxia (SARA), score range 0-40, higher score indicates higher ataxia severity
Measure of the usability of the program and hardware | Week 24
  Measured with the French System Usability Scale (F-SUS), original score range 0-40 converted to 0-100, a SUS score above a 68 would be considered above average and anything below 68 is below average
Change in sleep components | Week 12, week 24
  The sleep components are measured with an actigraphy watch
Change in mobility components | Week 12, week 24
  The changes in mobility components are measured with an actigraphy watch
Change in the adductor hip muscle group spasticity | Baseline, week 12, week 24
  Change in the adductor hip muscle group spasticity, measured with the Modified Ashworth Scale
Change in the knee extensor muscle group spasticity | Baseline, week 12, week 24
  Change in the knee extensor muscle group spasticity, measured with the Modified Ashworth Scale
Change in the knee flexor muscle group spasticity | Baseline, week 12, week 24
  Change in the knee flexor muscle group spasticity, measured with the Modified Ashworth Scale
Change in the plantar flexor muscle group spasticity | Baseline, week 12, week 24
  Change in the plantar flexor muscle group spasticity, measured with the Modified Ashworth Scale
Sum of lower limb muscle spasticity | Baseline, week 12, week 24
  Sum of the spasticity results obtained for the adductor hip, knee extensor, knee flexor and plantar flexor muscle groups

CONTACTS AND LOCATIONS:
Overall Officials: Elise Duchesne, Ph.D, Principal Investigator — Université du Québec à Chicoutimi
Locations (1):
- Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Saguenay, Quebec, Canada